CLINICAL TRIAL: NCT04357691
Title: Effects of Different Cardiorespiratory Training Program on Endurance Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wang Yongtai Raymond (Other)
Collaborators: The N.1 Institute for Health (N.1) (Other)
Responsible Party: Sponsor-Investigator, Wang Yongtai Raymond, Research Associate, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Project CURATE
Record Dates: First submitted 2020-04-07; First posted 2020-04-22 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy individuals (low-high-mod) (Other): Participants will undergo the calibration phase beginning with low intensity training, followed by high, and moderate intensity training. Each training intensity will be performed 3 days a week for 2 weeks
  Interventions: Behavioral: Conventional training; Behavioral: AI-led training
- Healthy individuals (mod-high-low) (Other): Participants will undergo the calibration phase beginning with moderate intensity training, followed by high, and low intensity training. Each training intensity will be performed 3 days a week for 2 weeks
  Interventions: Behavioral: Conventional training; Behavioral: AI-led training
- Healthy individuals (mod-low-high) (Other): Participants will undergo the calibration phase beginning with moderate intensity training, followed by low, and high intensity training. Each training intensity will be performed 3 days a week for 2 weeks.
  Interventions: Behavioral: Conventional training; Behavioral: AI-led training

INTERVENTIONS:
Behavioral: Conventional training — Participants will perform a conventional training for 4 weeks, using low-moderate-high-low intensity progression training model
Behavioral: AI-led training — Participants will perform an AI-led training for 4 weeks

SUMMARY:
Conventional training methods are typically administered in a fixed progressive manner, which can lead to sub-optimal responses and injuries. Artificial intelligence (i.e. CURATE.AI) can be harnessed to personalise physical training strategies. Using a single participant training profile, a parabolic/quadratic response to the intervention can be generated to identify the training intensity needed to optimise training outcomes. Previous studies showed CURATE.AI could dynamically modulate drug dosing in oncology. Extending the utility of results to human performance, this study will adapt CURATE.AI with the goal of optimising endurance performance through individualised training regimes.

Up to 20 participants will be recruited and randomised into two groups to undergo a calibration phase, which involves performing 3 sessions of exercise sessions per week over 2 weeks per intensity (low, moderate and high) in a crossover study design. Exercise sessions will be interspersed with a 2.4 km time trial, a VO2peak test and 2 weeks of wash out period. The utility phase will divide participants into two groups to undergo 3 exercise sessions per week, totalling to 12 exercise sessions. Either an AI-led training or a conventional training programme will be performed to compare the differences in training outcomes. Blood plasma will be obtained at selected time points in both phases to evaluate the effects of training on blood lipid profiles.

Findings from this study can potentially optimise efficacy and efficiency of endurance performance through personalised training with AI.

DETAILED DESCRIPTION:
Participants:

Up to 20 recreationally active healthy males, aged between 21 to 35 years, will be recruited to take part in this study. All volunteers will provide their informed consent in writing before participating in the study. The possible risk and benefits will be made known to the participant prior to the agreement to participate and they will be allowed to withdraw from the study at any point in time without any reason provided. All potential participants will first be required to undergo medical screening by a certified independent practitioner before participating in the study. The medical practitioner conducting the assessment will be informed of the purpose of the medical screening. The screening is to ensure that the potential participant is eligible to take part in the study. The personal particulars form will also be completed by each participant prior to the commencement of each trial.

Baseline measurements and familiarisation trials:

In the first session, anthropometry measurements will be taken. Based on the height and nude body mass, the body mass index (BMI) will be calculated (body mass in kg) / (height in m)2. Waist and hip circumference will be determined using a measuring tape. Skinfold thickness measurements will be taken at 4 sites (biceps, triceps, subscapular and suprailiac) in triplicate using skinfold calliper and the mean value will be used to calculate total skin fold. Body density will be calculated according to the estimation of Durnin and Womersley (1974) and percentage body fat will be estimated using the equation of Siri (1956).

Familiarisation of the 2.4 km time trial and the treadmill peak oxygen uptake (VO2peak) test will be performed 2 weeks before the commencement of the actual 2.4 km time trial. Ample rest is given between the two sessions for recovery.

Control of trial status:

Before the commencement of every trials, participants will be reminded to remain hydrated by consuming sufficient fluids, to have at least 8 hours of sleep, to refrain from alcoholic beverages, and to refrain from any forms of strenuous physical activity 24 h before each trial. Blood glucose will be measured before the start of the session via finger pricked using a lancing device. Prior to the pricking of the finger, the site will be disinfected with an alcohol wipe(s) and pressure will be applied to the site of the prick after blood sampling to minimise any bruising that may develop. In addition, Participants will be required to perform a 2-day dietary record prior to every blood draw session. They will be requested to refrain from participating in other aerobic training regimes (other than the prescribed exercise routine) or any acute strenuous bout of exercise that is not part of their routine during the study period.

Study design:

Participants will be required to undergo endurance interval training with low, moderate or high intensity. Each training session will comprise a warm-up run (50-60% VO2peak) followed by a 1-min fast run (80 to 140% VO2peak) interspersed with 1-min of recovery between each running bout till participants reach 18 out of 20 on the ratings of perceived exertion (RPE; Borg's scale). Participants will perform 10-15 repetitions of interval runs during each session. Heart rate, RPE, and blood pressure will be measured continuously at stipulated intervals. Water will be provided ad libitum during all training sessions. In the utility phase, participants will either perform an AI-led training or a conventional training program for 4 weeks. A 2.4 km time trial and a treadmill peak oxygen uptake (VO2peak) test will be conducted at baseline, in between the low, moderate and high intensity bouts of training in the calibration phase, and before the first and last week of the utility phase. Similar to the familiarisation trials, the treadmill VO2peak test and 2.4 km time trial will be done at 3 days apart from each other to allow for recovery. The two phases would consist of 47 sessions, inclusive of seven VO2peak tests and seven 2.4 km time trials. The total duration for each participant will take approximately 6 months.

Blood sampling and analysis:

After 5 min of seated rest, participant will immerse their arm in warm water (42-45°C) for 10 min to promote arterialisation of venous blood. Blood (10 ml) will be withdrawn from the antecubital vein of the participants into an ETDA vacutainer tube for subsequent analysis of the lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Do not smoke or use tobacco products (including shisha)
* BMI < 30
* Medically fit
* 2.4 km run time of 10 to 14 minutes in the past 12 months

Exclusion Criteria:

•Individuals with a history of existing musculoskeletal injury or respiratory diseases

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in 2.4 km completion time following first cycle in phase 1 | Baseline and Week 4 of phase 1 (phase 1 first cycle consist of 42 days)
  Time taken to complete 2.4 km
Changes in 2.4 km completion time following second cycle in phase 1 | Baseline and Week 9 of phase 1 (phase 1 second cycle consist of 35 days)
  Time taken to complete 2.4 km
Changes in 2.4 km completion time following third cycle in phase 1 | Baseline and Week 14 of phase 1 (phase 1 third cycle consist of 21 days)
  Time taken to complete 2.4 km
Changes in 2.4 km completion time following phase 2 | Baseline and Week 6 of phase 2 (phase 2 consist of 49 days)
  Time taken to complete 2.4 km

SECONDARY OUTCOMES:
Changes in VO2peak following first cycle in phase 1 | Baseline and Week 4 of phase 1 (phase 1 first cycle consist of 42 days)
  Measurement of oxygen uptake under maximal work capacity
Changes in VO2peak following second cycle in phase 1 | Baseline and Week 9 of phase 1 (phase 1 second cycle consist of 35 days)
  Measurement of oxygen uptake under maximal work capacity
Changes in VO2peak following third cycle in phase 1 | Baseline and Week 14 of phase 1 (phase 1 third cycle consist of 21 days)
  Measurement of oxygen uptake under maximal work capacity
Changes in VO2peak following phase 2 | Baseline and Week 6 of phase 2 (phase 2 consist of 49 days)
  Measurement of oxygen uptake under maximal work capacity
Resting blood lipids panel (triglycerides, cholesterols, phospholipids, sphingolipids, inflammatory lipids, testosterone, cortisol, endocannabinoids) in phase 1 | Week 1 of phase 1 (phase 1 consist of 98 days)
  Lipid biomarkers related to metabolism, inflammation, fitness, health, and pain
Changes in blood lipids panel (triglycerides, cholesterols, phospholipids, sphingolipids, inflammatory lipids, testosterone, cortisol, endocannabinoids) pre- and post- training following first cycle in phase 1 | Week 2 and 3 of phase 1 (phase 1 first cycle consist of 42 days)
  Lipid biomarkers related to metabolism, inflammation, fitness, health, and pain
Changes in blood lipids panel (triglycerides, cholesterols, phospholipids, sphingolipids, inflammatory lipids, testosterone, cortisol, endocannabinoids) pre- and post- training following second cycle in phase 1 | Week 7 and 8 of phase 1 (phase 1 second cycle consist of 35 days)
  Lipid biomarkers related to metabolism, inflammation, fitness, health, and pain
Changes in blood lipids panel (triglycerides, cholesterols, phospholipids, sphingolipids, inflammatory lipids, testosterone, cortisol, endocannabinoids) pre- and post- training following third cycle in phase 1 | Week 12 and 13 of phase 1 (phase 1 third cycle consist of 21 days)
  Lipid biomarkers related to metabolism, inflammation, fitness, health, and pain
Changes in resting blood lipids panel (triglycerides, cholesterols, phospholipids, sphingolipids, inflammatory lipids, testosterone, cortisol, endocannabinoids) in phase 2 | Week 1 and 7 of phase 2 (phase 2 consist of 49 days)
  Lipid biomarkers related to metabolism, inflammation, fitness, health, and pain
Changes in blood lipids panel (triglycerides, cholesterols, phospholipids, sphingolipids, inflammatory lipids, testosterone, cortisol, endocannabinoids) pre- and post- training in phase 2 | Week 2, 4 and 5 of phase 2 (phase 2 consist of 49 days)
  Lipid biomarkers related to metabolism, inflammation, fitness, health, and pain

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wei, Jason Lee, PhD, Principal Investigator — National University of Singapore; Dean Ho, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
This is in compliance with the national personal data protection act. Institutions would need to abide to the data protection law when handling personal data. However, ample information has been provided in the inclusion and exclusion criteria to understand the participant's demographics used in this study.

REFERENCES:
- [Background] Wang H, Lee DK, Chen KY, Chen JY, Zhang K, Silva A, Ho CM, Ho D. Mechanism-independent optimization of combinatorial nanodiamond and unmodified drug delivery using a phenotypically driven platform technology. ACS Nano. 2015 Mar 24;9(3):3332-44. doi: 10.1021/acsnano.5b00638. Epub 2015 Feb 23. PMID 25689511
- [Background] Rashid MBMA, Toh TB, Hooi L, Silva A, Zhang Y, Tan PF, Teh AL, Karnani N, Jha S, Ho CM, Chng WJ, Ho D, Chow EK. Optimizing drug combinations against multiple myeloma using a quadratic phenotypic optimization platform (QPOP). Sci Transl Med. 2018 Aug 8;10(453):eaan0941. doi: 10.1126/scitranslmed.aan0941. PMID 30089632